CLINICAL TRIAL: NCT02325752
Title: A Prospective Randomised Control Trial to Study the Effectiveness of a Health Service Innovation Using a Modified Virtual Ward Model to Prevent Unscheduled Readmission of High Risk Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Agency for Integrated Care, Singapore (Other); Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2011/380/E
Record Dates: First submitted 2014-12-21; First posted 2014-12-25 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Chronic Diseases
Keywords: readmission; chronic diseases
MeSH Terms: conditions — Chronic Disease | interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Patients in the control group received usual care by the hospital. There was no contact between the patients in the control group and the study team throughout the 3 months interval. A scheduled telephone call was made at the end of 3 months when they were invited to participate in a telephone survey.
- Intervention (Active Comparator): Intervention
  Interventions: Other: Intervention

INTERVENTIONS:
Other: Intervention — A multidisciplinary team delivered the transitional care program.
  Our transitional care program focused on four key areas:
  1. Post discharge surveillance of the patient to ensure adherence to care plans.
  2. Coordination of follow-up visits with specialist care providers.
  3. Patent education and care giver training.
  4. Activation of community and social services.
  Upon recruitment, the patients were interviewed and assessed by the team nurse prior to their discharge. Intervention starts upon discharge from the hospital. The duration of the intervention program was 3 months. A follow-up by telephone was made within 72 hours after discharge to assess patient's condition and adherence to treatment plan. Home visits were made within 2 weeks after discharge.
  Arms: Intervention

SUMMARY:
The investigators conducted an open randomized control study of patients who received the transitional care program versus patients who received usual care at the Singapore General Hospital from Aug 2011 to Sept 2012.

DETAILED DESCRIPTION:
The investigators conducted an open randomized control study of patients who received the transitional care program versus patients who received usual care at the Singapore General Hospital from Aug 2011 to Sept 2012.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 2 or more unscheduled admission in the last 90 days to selected medical departments
* LACE score of ≥10.

Exclusion Criteria:

* Non-residents
* No telephone contact or a resident address
* Residing in long term care facilities.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 840 (Actual)
Dates: Start 2011-08; Primary Completion 2012-10 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Rate of readmission | 30 days
  Any hospital admission after randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Kheng Hock Lee, MBBS, Principal Investigator — Singhealth Foundation

REFERENCES:
- [Derived] Lee KH, Low LL, Allen J, Barbier S, Ng LB, Ng MJ, Tay WY, Tan SY. Transitional care for the highest risk patients: findings of a randomised control study. Int J Integr Care. 2015 Oct 22;15:e039. doi: 10.5334/ijic.2003. eCollection 2015 Oct-Dec. PMID 27118956